CLINICAL TRIAL: NCT02041091
Title: Pharmacokinetic Evaluations of Tabalumab Following Subcutaneous Administration by Prefilled Syringe or Auto Injector in Patients With Systemic Lupus Erythematosus
Brief Title: A Study of Tabalumab (LY2127399) Using Two Different Injection Methods in Participants With Lupus
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Lack of efficacy
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15193; H9B-MC-BCEI (Other: Eli Lilly and Company)
Record Dates: First submitted 2014-01-17; First posted 2014-01-20 (Estimated); Results first posted 2018-06-15 (Actual); Last update posted 2018-06-15 (Actual); Status verified 2018-05

CONDITIONS: Lupus Erythematosus, Systemic
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — tabalumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tabalumab Auto-Injector (Experimental): Tabalumab given Week 0 as a loading dose of 240 milligram (mg) given as two subcutaneous (SC) injections each of 120 mg followed by 120 mg SC injection every two weeks for 12 weeks. Participants may continue on this treatment regimen for 52 weeks.
  Interventions: Drug: Tabalumab Auto-Injector
- Tabalumab Prefilled Syringe (Experimental): Tabalumab given Week 0 as a loading dose of 240 mg given as two SC injections each of 120 mg followed by 120 mg SC injections every two weeks for 12 weeks. Participants may continue to on this treatment regimen for 52 weeks.
  Interventions: Drug: Tabalumab Prefilled Syringe

INTERVENTIONS:
Drug: Tabalumab Auto-Injector — Administered SC
  Other Names: LY2127399
  Arms: Tabalumab Auto-Injector
Drug: Tabalumab Prefilled Syringe — Administered SC
  Other Names: LY2127399
  Arms: Tabalumab Prefilled Syringe

SUMMARY:
The purpose of this study is to evaluate the amount of tabalumab in the blood after it is given by two different injection methods - A traditional syringe or a spring loaded syringe for 12 weeks. Participants may continue to receive study drug for up to 52 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Lupus.
* Able and willing to have blood drawn for PK sampling.

Exclusion Criteria:

* Have severe active lupus nephritis.
* Have severe active central nervous system (CNS) or peripheral neurologic disease or other severe neurologic involvement requiring treatment within approximately 3 months prior to screening.
* Have received high dose corticosteroid within approximately 1 month prior to baseline.
* Have initiated or adjusted treatment with immunosuppressant drugs within approximately 1 month prior to baseline.
* Have received plasmapheresis within approximately 3 months prior to baseline.
* Have previously received approved or experimental B cell targeted therapies within the last year.
* Have received any biologic or non-biologic therapy within approximately 3 months or 5 half-lives (whichever is longer).
* Have a history of severe reaction to any biologic therapy.
* Have an active or recent infection within approximately 1 month prior to Week 0.
* Have had a serious infection within approximately 3 month or serious bone/joint infection within approximately 6 months prior to baseline.
* Have evidence of or test positive for active hepatitis B or are positive for hepatitis C or human immunodeficiency virus (HIV).
* Have evidence of active or latent tuberculosis.
* Have significant hematological abnormalities.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 226 (Actual)
Dates: Start 2014-01; Primary Completion 2014-10 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (44):
- United States (36):
  - Medvin Clinical Research, Covina, California
  - TriWest Research Associates, El Cajon, California
  - ProHealth Partners Medical Group, Long Beach, California
  - Wallace Rheumatic Study Center, Los Angeles, California
  - Desert Medical Advances, Palm Desert, California
  - Inlande Rheumatology Clinical Trials, Upland, California
  - Denver Arthritis Center, Denver, Colorado
  - New England Research Associates, Trumbull, Connecticut
  - Advanced Pharma Clinical Research, Miami, Florida
  - New Horizon Research Center, Miami, Florida
  - Arthritis Research of Florida, Palm Harbor, Florida
  - Clinical Research of West Florida, Inc., Tampa, Florida
  - Indiana University Health, Indianapolis, Indiana
  - The Arthritis & Diabetes Clinic Inc., Monroe, Louisiana
  - West Michigan Rheumatology, Grand Rapids, Michigan
  - Clayton Medical Research, St Louis, Missouri
  - Physician Research Collaboration, LLC, Lincoln, Nebraska
  - Westroads Clinical Research-Omaha, Omaha, Nebraska
  - Innovative Health Research, Las Vegas, Nevada
  - (AOA) Arthritis & Osteoporosis Associates, Freehold, New Jersey
  - Albuquerque Clinical Trials, Albuquerque, New Mexico
  - The Feinstein Institute for Medical Research, Manhasset, New York
  - Box Arthritis & Rheumatology of the Carolinas, PLLC, Charlotte, North Carolina
  - PharmQuest, Greensboro, North Carolina
  - Shanahan Rheumatology & Immunotherapy, Raleigh, North Carolina
  - PMG Research of Salisbury, Salisbury, North Carolina
  - Paramount Medical Research, Middleburg Heights, Ohio
  - Oklahoma Arthritis Center, Edmond, Oklahoma
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - Clinical Research Center of Reading, LLP, Wyomissing, Pennsylvania
  - Low Country Research Center, North Charleston, South Carolina
  - Tekton Research, Inc., Austin, Texas
  - Sun Research Institute, San Antonio, Texas
  - Virginia Clinical Research, Norfolk, Virginia
  - Arthritis Northwest Rheumatology, Spokane, Washington
  - Mountain State Clinical Research, Clarksburg, West Virginia
- Puerto Rico (5):
  - Office: Perez de Jesus, Amarylis, Caguas
  - Ramon L. Ortega Colon, Carolina
  - GCM Medical Group PSC, San Juan
  - Mindful Medical Research, San Juan
  - Latin Clinical Trial Center, Santurce
- South Korea (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Daejeon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Incheon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Seoul

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants who complete the Treatment Period will have the option of participating in the Optional Safety Extension Period through Week 52.
Groups:
- Tabalumab Prefilled Syringe: Tabalumab given Week 0 as a loading dose of 240 milligram (mg) given as two subcutaneous (SC) injections each of 120 mg followed by 120 mg SC injections every two weeks for 12 weeks. Participants may continue to on this treatment regimen for 52 weeks.
  The treatment regimen from Week 12 to Week 52 is an Optional Safety Extension Period.
  All participants will participate in a Post-Treatment Follow-Up Period regardless of their participation in the Optional Safety Extension Period.
- Tabalumab Auto-Injector: Tabalumab given Week 0 as a loading dose of 240 mg given as two SC injections each of 120 mg followed by 120 mg SC injection every two weeks for 12 weeks. Participants may continue on this treatment regimen for 52 weeks.
  The treatment regimen from Week 12 to Week 52 is an Optional Safety Extension Period.
  All participants will participate in a Post-Treatment Follow-Up Period regardless of their participation in the Optional Safety Extension Period.
Period: Treatment
Arm/Group | Tabalumab Prefilled Syringe | Tabalumab Auto-Injector
Started | 112 | 114
Received At Least One Dose of Study Drug | 112 | 114
Participated in Follow Up | 106 | 96
Completed | 90 | 91
Not Completed | 22 | 23
Not completed — Adverse Event | 3 | 3
Not completed — Withdrawal by Subject | 2 | 4
Not completed — Physician Decision | 1 | 0
Not completed — Sponsor Decision | 15 | 16
Not completed — Lost to Follow-up | 1 | 0
Period: Optional Safety Extension Period
Arm/Group | Tabalumab Prefilled Syringe | Tabalumab Auto-Injector
Started | 85 (Participation was optional for the Safety Extension Period.) | 82 (Participation was optional for the Safety Extension Period.)
Completed | 0 | 0
Not Completed | 85 | 82
Not completed — Adverse Event | 4 | 2
Not completed — Withdrawal by Subject | 5 | 2
Not completed — Protocol Violation | 2 | 0
Not completed — Physician Decision | 2 | 1
Not completed — Sponsor Decision | 70 | 74
Not completed — Lost to Follow-up | 2 | 3

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Tabalumab Prefilled Syringe | Tabalumab Auto-Injector | Total
Number analyzed (Participants) | 112 | 114 | 226
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.03 (12.691) | 44.93 (13.306) | 45.97 (13.018)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 106 | 108 | 214
  Male | 6 | 6 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 26 | 32 | 58
  Not Hispanic or Latino | 84 | 80 | 164
  Unknown or Not Reported | 2 | 2 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 15 | 13 | 28
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 15 | 22 | 37
  White | 82 | 76 | 158
  More than one race | 0 | 3 | 3
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 99 | 101 | 200
  South Korea | 13 | 13 | 26

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics (PK): Maximum Concentration (Cmax) of Tabalumab After Loading Dose
Description: Maximum serum concentration of tabalumab, after the loading dose, assessed over the 14-day dosing interval, stratified by device.PK samples taken during the first dosing interval, days 4, 7, 9, 11, 14, were analyzed using noncompartmental analysis (NCA) methods to calculate the geometric mean.
Time Frame: Day 4, 7, 9, 11, 14: collected at approximately the same time of day as the administration of the Week 0 injection of tabalumab
Population: PK population: all randomized participants who received at least one dose of the study drug and had evaluable tabalumab PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram per milliliter (ug/mL)
Arm/Group | Tabalumab Prefilled Syringe | Tabalumab Auto-Injector
Number analyzed (Participants) | 87 | 99
microgram per milliliter (ug/mL) | 35.7 (53.2) | 34.1 (46.5)

2. Primary Outcome: Pharmacokinetics (PK): Area Under the Concentration Time Curve From Time 0 to 14 Days (AUC 0-14) of Tabalumab After Loading Dose
Description: Area under the concentration time curve after the loading dose, assessed over the 14-day dosing interval, stratified by device.PK samples taken during the first dosing interval, days 4, 7, 9, 11, 14, were analyzed using NCA methods to calculate the geometric mean.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram*hour per milliliter (ug*hr/mL)
Arm/Group | Tabalumab Prefilled Syringe | Tabalumab Auto-Injector
Number analyzed (Participants) | 87 | 99
microgram*hour per milliliter (ug*hr/mL) | 8390 (44.0) | 8170 (41.3)

3. Secondary Outcome: Pharmacokinetics (PK): Cmax of Tabalumab Based on Body Weight
Description: Maximum serum concentration of tabalumab, after the loading dose, assessed over the 14-day dosing interval , stratified by body weight (low <60 kilograms (kg), medium 60kg- 100kg, high >100kg).PK samples taken during the first dosing interval, days 4, 7, 9, 11, 14, were analyzed using NCA methods to calculate the geometric mean.
Time Frame: as for outcome 1
Population: PK population: all randomized participants who received at least one dose of the study drug and had evaluable tabalumab PK data. The analyses was conducted on tabalumab exposure parameter from both arms combined per the statistical analysis plan, since the tabalumab exposure was similar following prefilled syringe and auto-injector injections.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/mL
Groups:
- Total PK Population: Total participants randomized to prefilled syringe or auto-injector arm from randomization through week 61.
Arm/Group | Total PK Population
Number analyzed (Participants) | 186
μg/mL
  Low: number analyzed (Participants) | 62
  Low | 47.8 (40.5)
  Medium: number analyzed (Participants) | 63
  Medium | 34.7 (42.5)
  High: number analyzed (Participants) | 61
  High | 25.4 (40.1)

4. Secondary Outcome: Pharmacokinetics (PK): AUC 0-14 of Tabalumab Based on Body Weight
Description: Area under the concentration time curve after the loading dose, assessed over the 14-day dosing interval, stratified by body weight (low <60 kilograms (kg), medium 60kg- 100kg, high >100kg). PK samples taken during the first dosing interval, days 4, 7, 9, 11, 14, were analyzed using noncompartmental analysis (NCA) methods to calculate the geometric mean.
Time Frame: as for outcome 1
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug*hr/mL
Arm/Group | Total PK Population
Number analyzed (Participants) | 186
ug*hr/mL
  Low: number analyzed (Participants) | 62
  Low | 10800 (31.9)
  Medium: number analyzed (Participants) | 63
  Medium | 8450 (35.5)
  High: number analyzed (Participants) | 61
  High | 6160 (36.7)

5. Secondary Outcome: Number of Participants Reporting Incomplete Tabalumab Dose Administration
Description: Participants reporting incomplete dose administration from the study drug administration log.
Time Frame: Week 0 through Week 12
Population: Safety population: all randomized patients who received at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Tabalumab Prefilled Syringe | Tabalumab Auto-Injector
Number analyzed (Participants) | 112 | 114
Participants | 0 | 1

6. Secondary Outcome: Number of Participants Developing Anti-Tabalumab Antibodies
Description: Participants with treatment-emergent anti-tabalumab antibodies were participants who had any samples from baseline up to and through Week 12 that was a 4-fold increase (2-dilution increase) in immunogenicity titer over baseline titer, or participants who tested negative at baseline and positive post-baseline (at titer of ≥1:20). Baseline is defined as the last non-missing observation on or prior to the date of the first injection of tabalumab. Percentage of participants with anti-tabalumab antibodies = (number of participants with treatment-emergent anti-tabalumab antibodies / number of participants assessed)*100.
Time Frame: Week 0 through Week 12
Population: Safety population: all randomized participants who received at least 1 dose of study treatment. Participants with a baseline sample and at least 1 evaluable sample after administration of study drug OR participants with no baseline sample and all evaluable post-baseline samples.
Measure: Count of Participants; unit: Participants
Arm/Group | Tabalumab Prefilled Syringe | Tabalumab Auto-Injector
Number analyzed (Participants) | 111 | 112
Participants | 1 | 0

7. Secondary Outcome: Subcutaneous Administration Assessment Questionnaire (SQAAQ) Score
Description: The SQAAQ is a 12-item questionnaire using a 7-point Likert scale (from "Strongly Disagree" as 1 to "Strongly Agree" as 7) that provides assessment of ease of use and confidence with using a prefilled syringe or auto-injector to administer a subcutaneous injection of drug. The 12 items are: A-Easy for me to learn how to use, B-Easy for me to unlock, C- Easy to hold in my hand when I inject my dose, D- Easy to inject my dose, E- Easy to know that my dose is complete, F- Easy to store the device in my refrigerator, G- Easy to remove needle shield/cover, H- Easy to pick up, I- Overall, easy to use, J- The device is stable against my skin during the injection, K- I am confident in my ability to use the device, L- I am confident my dose is complete.
Time Frame: Week 0, Week 4 and Week 8
Population: Safety population: all randomized patients who received at least 1 dose of study treatment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tabalumab Prefilled Syringe | Tabalumab Auto-Injector
Number analyzed (Participants) | 112 | 114
units on a scale
  Week 0: A | 6.5 (1.14) | 6.8 (0.60)
  Week 0: B: number analyzed (Participants) | 107 | 114
  Week 0: B | 5.9 (1.39) | 6.8 (0.60)
  Week 0: C | 6.3 (1.24) | 6.8 (0.55)
  Week 0: D | 6.4 (1.12) | 6.8 (0.45)
  Week 0: E | 6.5 (0.92) | 6.7 (0.56)
  Week 0: F: number analyzed (Participants) | 112 | 113
  Week 0: F | 6.6 (0.82) | 6.7 (0.70)
  Week 0: G | 6.3 (1.31) | 6.5 (0.74)
  Week 0: H | 6.6 (0.82) | 6.9 (0.35)
  Week 0: I | 6.4 (1.06) | 6.9 (0.39)
  Week 0: J | 6.4 (1.12) | 6.8 (0.47)
  Week 0: K | 6.6 (0.93) | 6.9 (0.40)
  Week 0: L | 6.7 (0.81) | 6.8 (0.51)
  Week 4: A: number analyzed (Participants) | 95 | 110
  Week 4: A | 6.7 (0.59) | 6.8 (0.71)
  Week 4: B: number analyzed (Participants) | 93 | 110
  Week 4: B | 6.4 (0.94) | 6.8 (0.64)
  Week 4: C: number analyzed (Participants) | 95 | 110
  Week 4: C | 6.5 (0.97) | 6.8 (0.71)
  Week 4: D: number analyzed (Participants) | 95 | 110
  Week 4: D | 6.5 (0.97) | 6.8 (0.73)
  Week 4: E: number analyzed (Participants) | 95 | 110
  Week 4: E | 6.5 (0.95) | 6.7 (0.76)
  Week 4: F: number analyzed (Participants) | 95 | 110
  Week 4: F | 6.6 (0.84) | 6.8 (0.73)
  Week 4: G: number analyzed (Participants) | 95 | 110
  Week 4: G | 6.5 (0.77) | 6.5 (1.05)
  Week 4: H: number analyzed (Participants) | 95 | 110
  Week 4: H | 6.7 (0.59) | 6.8 (0.64)
  Week 4: I: number analyzed (Participants) | 95 | 110
  Week 4: I | 6.5 (0.87) | 6.8 (0.70)
  Week 4: J: number analyzed (Participants) | 95 | 110
  Week 4: J | 6.5 (0.92) | 6.7 (0.78)
  Week 4: K: number analyzed (Participants) | 95 | 110
  Week 4: K | 6.6 (0.68) | 6.8 (0.65)
  Week 4: L: number analyzed (Participants) | 95 | 110
  Week 4: L | 6.7 (0.82) | 6.8 (0.77)
  Week 8: A: number analyzed (Participants) | 88 | 94
  Week 8: A | 6.7 (0.58) | 6.9 (0.30)
  Week 8: B: number analyzed (Participants) | 88 | 94
  Week 8: B | 6.5 (1.07) | 6.9 (0.28)
  Week 8: C: number analyzed (Participants) | 88 | 94
  Week 8: C | 6.6 (0.86) | 6.9 (0.37)
  Week 8: D: number analyzed (Participants) | 88 | 94
  Week 8: D | 6.6 (0.96) | 6.9 (0.31)
  Week 8: E: number analyzed (Participants) | 88 | 94
  Week 8: E | 6.6 (0.86) | 6.8 (0.74)
  Week 8: F: number analyzed (Participants) | 88 | 94
  Week 8: F | 6.8 (0.73) | 6.8 (0.74)
  Week 8: G: number analyzed (Participants) | 88 | 94
  Week 8: G | 6.6 (0.89) | 6.6 (1.06)
  Week 8: H: number analyzed (Participants) | 88 | 94
  Week 8: H | 6.8 (0.48) | 6.8 (0.68)
  Week 8: I: number analyzed (Participants) | 88 | 94
  Week 8: I | 6.7 (0.81) | 6.9 (0.67)
  Week 8: J: number analyzed (Participants) | 88 | 94
  Week 8: J | 6.6 (1.03) | 6.8 (0.74)
  Week 8: K: number analyzed (Participants) | 88 | 94
  Week 8: K | 6.7 (0.82) | 6.9 (0.67)
  Week 8: L: number analyzed (Participants) | 88 | 94
  Week 8: L | 6.8 (0.58) | 6.8 (0.72)

8. Secondary Outcome: Pharmacokinetics (PK): Cmax of Tabalumab Based on Injection Site Stratifications
Description: Maximum serum concentration of tabalumab in medium body weight group, after the loading dose via auto-injector, assessed over the 14-day dosing interval, stratified by injection site. PK samples taken during the first dosing interval, days 4, 7, 9, 11, 14, were analyzed using noncompartmental analysis (NCA) methods to calculate the geometric mean.
Time Frame: as for outcome 1
Population: PK population (all randomized participants who received at least one dose of the study drug and had evaluable tabalumab PK data) in medium body weight group, dosed by auto-injector.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/mL
Arm/Group | Tabalumab Auto-Injector
Number analyzed (Participants) | 33
μg/mL
  Arm: number analyzed (Participants) | 21
  Arm | 29.4 (38.1)
  Abdomen: number analyzed (Participants) | 19
  Abdomen | 37 (35.4)
  Thigh: number analyzed (Participants) | 23
  Thigh | 42.2 (52.6)

9. Secondary Outcome: Pharmacokinetics (PK): AUC 0-14 of Tabalumab Based on Injection Site Stratifications
Description: Area under the concentration time curve in medium body weight group after the loading dose via auto-injector, assessed over the 14-day dosing interval, stratified by injection site. PK samples taken during the first dosing interval, days 4, 7, 9, 11, 14, were analyzed using noncompartmental analysis (NCA) methods to calculate the geometric mean.
Time Frame: as for outcome 1
Population: as for outcome 8
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg*hr/mL
Arm/Group | Tabalumab Auto-Injector
Number analyzed (Participants) | 33
μg*hr/mL
  Arm: number analyzed (Participants) | 21
  Arm | 7380 (36)
  Abdomen: number analyzed (Participants) | 19
  Abdomen | 8890 (27.9)
  Thigh: number analyzed (Participants) | 23
  Thigh | 10000 (34)

ADVERSE EVENTS:
Description: All participants who received at least 1 dose of study drug.
Groups:
- Tabalumab Prefilled Syringe Treatment: Tabalumab given Week 0 as a loading dose of 240 mg given as two SC injections each of 120 mg followed by 120 mg SC injections every two weeks for 12 weeks.
- Tabalumab Auto-Injector Treatment: Tabalumab given Week 0 as a loading dose of 240 mg given as two SC injections each of 120 mg followed by 120 mg SC injection every two weeks for 12 weeks.
- Prefilled Syringe Optional Safety Extension: Tabalumab given SC every two weeks from Week 12 to Week 52.
- Auto-Injector Optional Safety Extension: Tabalumab given every two weeks from Week 12 to Week 52.
- Prefilled Syringe Follow Up; Auto-Injector Follow Up: Follow Up 24-48 weeks post last doseTabalumab
Arm/Group | Tabalumab Prefilled Syringe Treatment | Tabalumab Auto-Injector Treatment | Prefilled Syringe Optional Safety Extension | Auto-Injector Optional Safety Extension | Prefilled Syringe Follow Up | Auto-Injector Follow Up
Serious Adverse Events (participants affected / at risk) | 1/112 | 1/114 | 1/85 | 2/82 | 4/106 | 8/96
Other Adverse Events (participants affected / at risk) | 79/112 | 65/114 | 37/85 | 25/82 | 7/106 | 15/96
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Tabalumab Prefilled Syringe Treatment (N=112) | Tabalumab Auto-Injector Treatment (N=114) | Prefilled Syringe Optional Safety Extension (N=85) | Auto-Injector Optional Safety Extension (N=82) | Prefilled Syringe Follow Up (N=106) | Auto-Injector Follow Up (N=96)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sideropenic dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cholecystitis chronic (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gallbladder cholesterolosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hepatic steatosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tracheobronchitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ear infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Appendicitis perforated (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Major depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Suicide attempt (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Major depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Suicide attempt (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Renal cyst (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Menorrhagia (Reproductive system and breast disorders) | 0/106 (0) | 1/108 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0/81 (0) | 1/79 (1) | 0 (0) | 0 (0)
Haemorrhagic ovarian cyst (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1/100 (1) | 0/90 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Peripheral artery bypass (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral arterial occlusive disease (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tabalumab Prefilled Syringe Treatment (N=112) | Tabalumab Auto-Injector Treatment (N=114) | Prefilled Syringe Optional Safety Extension (N=85) | Auto-Injector Optional Safety Extension (N=82) | Prefilled Syringe Follow Up (N=106) | Auto-Injector Follow Up (N=96)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 5 (6) | 5 (8) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 7 (7) | 4 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site bruising (General disorders) | 3 (4) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site erythema (General disorders) | 4 (6) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site pain (General disorders) | 4 (5) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site pruritus (General disorders) | 3 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site reaction (General disorders) | 8 (19) | 14 (37) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site swelling (General disorders) | 5 (7) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Local swelling (General disorders) | 2 (2) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site erythema (General disorders) | 0 (0) | 0 (0) | 2 (3) | 1 (3) | 0 (0) | 0 (0)
Injection site pruritus (General disorders) | 0 (0) | 0 (0) | 2 (4) | 0 (0) | 0 (0) | 0 (0)
Injection site reaction (General disorders) | 0 (0) | 0 (0) | 4 (8) | 8 (16) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 6 (7) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 2 (2) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 5 (6) | 5 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (5)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 5 (6)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Cardiac murmur (Investigations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (6) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 3 (4) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 6 (7) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 2 (5) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 2 (3) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (4) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days